CLINICAL TRIAL: NCT00647192
Title: EPLERAF-Study: Eplerenone in the Prevention of Atrial Fibrillation Recurrences After Cardioversion
Acronym: EPLERAF
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Inclusion rate too low. Recruitment of further study centers too costly.
Sponsor: University Hospital, Saarland (Other)
Collaborators: University Medical Center Groningen (Other); Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: EPLERAF-01; Version 09_D; EudraCT number: 2007-002119-17
Record Dates: First submitted 2008-03-26; First posted 2008-03-31 (Estimated); Last update posted 2012-02-10 (Estimated); Status verified 2012-02

CONDITIONS: Atrial Fibrillation
Keywords: atrial fibrillation; electrical cardioversion; prevention of atrial fibrillation recurrence; mineralocorticoid receptor blocker; eplerenone; Recurrence of atrial fibrillation after cardioversion
MeSH Terms: conditions — Atrial Fibrillation | interventions — Eplerenone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Eplerenone treatment
  Interventions: Drug: Eplerenone
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Eplerenone — 50 mg per day
  Arms: 1
Drug: Placebo — 50 mg per day
  Arms: 2

SUMMARY:
The purpose of this study is to determine whether Eplerenone reduces atrial fibrillation (AF) recurrences within the first 8 weeks after electrical cardioversion of persistent AF.

ELIGIBILITY:
Inclusion Criteria:

* Persistent atrial fibrillation (AF), AF persistence for > 7 days but < 1 year
* Total AF history < 2 years
* Written informed consent of the patient
* Age ≥18 years
* Female patients are sterilised or postmenopausal or apply an adequate method for contraception (Pearl index <1%) and have a negative pregnancy test (ß-HCG) and do not breastfeed/nurse.

Exclusion Criteria:

* Hemodynamic instability or symptoms not allowing cardioversion to be delayed for 3 weeks
* Myocardial infarction within the last 3 months
* Heart failure NYHA class III - IV
* Uncontrolled hypertension, defined as a systolic blood pressure > 160 mm Hg and/or a diastolic blood pressure > 95 mm Hg (anti-hypertensive treatment is allowed).
* Pre-treatment with an aldosterone antagonist or other potassium sparing diuretics
* Instable angina pectoris
* Use of Digitalis
* Use of class I or class III antiarrhythmic drugs (must be stopped at least 5 half-life before)
* Contraindication or hypersensitivity to ß-blockers
* Open heart surgery within the last 3 months
* Pregnancy
* Acute and reversible illnesses
* Acute and chronic infection
* Alcohol or drug abuse or a severe progressive extracardiac disease
* Untreated manifest and latent hyper- or hypothyroidism or < 3 months peripheral euthyroidism (normal fT3)
* Moderate to severe renal insufficiency (Creatinine clearance less than 50 ml/min)
* Patients with liver cirrhosis (Child-Pugh class C)
* Co-administration of strong CYP3A4 inhibitors (e.g. Itraconazole, Ketoconazole, Ritonavir, Nelfinavir, Clarithromycin, Telithromycin and Nephazodon)
* Hypersensitivity against Eplerenone and/or one of the other components of the tablet (see Fachinformation)
* Serum potassium > 5 mmol/l
* Patients unlikely to comply with the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2008-03; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Atrial fibrillation recurrence after electrical cardioversion of atrial fibrillation | 8 weeks

SECONDARY OUTCOMES:
Sinus rhythm within eplerenone treatment before planned electrical cardioversion | 3 weeks
Cardioversion success | at least one sinus beat
Time to recurrence of atrial fibrillation | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Michael Böhm, MD, Principal Investigator — Universitätsklinikum des Saarlandes, Klinik für Innere Medizin III
Locations (2):
- Universitätsklinikum des Saarlandes, Klinik für Innere Medizin III, Homburg/Saar, Germany
- Rijksuniversiteit Groningen, Universitair Medisch Centrum, Groningen, Netherlands